CLINICAL TRIAL: NCT00597909
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Two Doses of AMMONUL® (Sodium Phenylacetate and Sodium Benzoate) Injection 10% / 10% in Subjects With Grade 3 or 4 Hepatic Encephalopathy
Brief Title: Efficacy and Safety Study of Ammonul® in Patients With Grade 3 or 4 Hepatic Encephalopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of enrollment and business decisions.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYP1203-004
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Encephalopathy
Keywords: Ammonul®; sodium phenylacetate and sodium benzoate; hepatic encephalopathy; Grade 3 or 4 Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy; Lymphoma, Follicular | interventions — phenylacetic acid; Sodium Benzoate; ammonul; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: sodium phenylacetate and sodium benzoate injection 10% / 10%
- Arm 2 (Experimental)
  Interventions: Drug: sodium phenylacetate and sodium benzoate injection 10% / 10%
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo solution (10% dextrose)

INTERVENTIONS:
Drug: sodium phenylacetate and sodium benzoate injection 10% / 10% — 5.5 g/m² diluted in 10% dextrose, IV as a 2-hour loading (initial) dose, followed by the same dose over 24 hours (maintenance infusion); maintenance infusion will be continued for 3 days (70 hours)
  Other Names: Ammonul®
  Arms: Arm 1
Drug: sodium phenylacetate and sodium benzoate injection 10% / 10% — 2.75 g/m² diluted in 10% dextrose, IV as a 2-hour loading (initial) dose, followed by the same dose over 24 hours (maintenance infusion); maintenance infusion will be continued for 3 days (70 hours)
  Other Names: Ammonul®
  Arms: Arm 2
Drug: placebo solution (10% dextrose) — Placebo solution (10% dextrose), IV as a 2-hour loading (initial) dose, followed by the same dose over 24 hours (maintenance infusion); maintenance infusion will be continued for 3 days (70 hours)
  Arms: Arm 3

SUMMARY:
The primary purpose of this study is to evaluate the safety and effectiveness of Ammonul® in subjects who become hospitalized with Grade 3 or 4 hepatic encephalopathy (HE).

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a reversible neuropsychiatric syndrome seen in patients with liver disease. The pathogenesis of HE is incompletely understood, but several pieces of evidence identify ammonia as a key factor in the development of HE. The liver normally detoxifies ammonia produced in the gastrointestinal tract. However, in patients with cirrhosis, portosystemic shunting allows ammonia to bypass the liver and reach the systemic circulation and the brain. The accumulation of ammonia in the brain, through mechanisms not yet fully defined, lead to changes of consciousness, intellectual function, and behavior.

Ammonul is currently approved as adjuvant therapy for the management of hyperammonemia and associated encephalopathy in patients with deficiencies in the enzymes of the urea cycle. Ammonul removes nitrogenous ammonia in these patients through pathways alternative to the urea cycle. It is anticipated that in patients with HE, Ammonul may lead to the scavenging of ammonia through these alternative biochemical pathways taking place in tissues other than the liver.

This study is designed to test the efficacy and safety of IV Ammonul® as a treatment for acute episodes of elevated ammonia in patients with Grade 3 or 4 HE. Study was terminated due to lack of enrollment and business decisions.

Study with completed results acquired from Horizon in 2024

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 75 years
* Signed written informed consent by subject's representative
* Current diagnosis of chronic liver disease with cirrhosis
* West Haven score of Grade 3 or 4 Hepatic Encephalopathy
* Weight between 45 and 150 kg
* Elevated venous ammonia concentration, defined as a value above the normal range at the local laboratory
* Estimated creatinine clearance of > 30 mL/min/1.73m², calculated using the Cockcroft-Gault formula, or serum creatinine < 2.5 mg/dL [Cockcroft-Gault formula: creatinine clearance = (140 - age) x weight in kg divided by (72 x serum creatinine in mg/dL); multiply result by 0.85 for females]
* Adequate urinary output of ≥ 30 mL/hour for the last 2 hours if estimated creatinine clearance is < 50 mL/min/1.73 m²
* Negative pregnancy test or documented sterilization procedure (tubal ligation or hysterectomy) or 5 years post-menopausal

Exclusion Criteria:

* Major gastrointestinal bleeding (hematemesis, melena, or hematochezia) requiring blood transfusion within the last 24 hours
* Uncontrolled sepsis, as defined by hemodynamic instability requiring vasopressor agents (renal-dosed dopamine allowed)
* Current diagnosis of acute hepatic failure
* Alcohol ingestion during last 24 hours
* Post liver transplant
* Serum sodium < 120 mEq/L
* Serum potassium ≤ 3.5 mEq/L
* Use of probenecid, valproate, penicillin or its derivatives, or corticosteroids (oral or IV) within the last 24 hours
* Use of any sedatives, benzodiazepines, or any neuro- or psycho-active drugs in the last 6 hours and a positive urinary drug screen
* Subjects who received any mind-altering agents (such as barbiturates, propofol, opioids, or benzodiazepines) to assist with intubation are not eligible while the effects of the drug are still apparent
* Congestive heart failure (New York Heart Association Class III or IV)
* Seizures, dementia, or any neurologic or psychiatric condition within the last 72 hours that may interfere with the assessment of the mental state
* Current diagnosis of major aspiration pneumonia or pulmonary edema accompanied by an oxygen saturation of ≤ 90% while breathing supplemental oxygen
* Laboratory test abnormalities determined to be clinically significant by the investigator
* Enrollment in another experimental (interventional) protocol within the last 30 days or 5 half-lives of the experimental drug, whichever s longer
* Any medical condition, which in the opinion of the investigator would constitute a contraindication to enrollment in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - UCSF-Fresno University, Fresno, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Permian Research Foundation, Odessa, Texas

REFERENCES:
- See also: Medline Plus: Brain Diseases — http://www.nlm.nih.gov/medlineplus/braindiseases.html
- See also: Medline Plus: Cirrhosis — http://www.nlm.nih.gov/medlineplus/cirrhosis.html
- See also: Medline Plus: Hepatitis — http://www.nlm.nih.gov/medlineplus/hepatitis.html
- See also: Medline Plus: Liver Diseases — http://www.nlm.nih.gov/medlineplus/liverdiseases.html
- See also: Medline Plus: Metabolic Disorders — http://www.nlm.nih.gov/medlineplus/metabolicdisorders.html
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled but did not receive drug or was randomized.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex/Gender, Customized [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, as Assessed by Time to Grade 2 or Less in the West Haven Criteria Sustaining for 4 Hours or Longer
Time Frame: Time to Grade 2 or less sustaining for 4 hours or longer
Population: One participant enrolled but did not receive drug or was randomized.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Safety, as Assessed by Reported Adverse Events, Clinical Laboratory Measurements, Changes in Vital Signs, and Changes in 12-lead ECG Results
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy, as Assessed by Proportion of Assessments With a 2-grade Improvement, Using West Haven Criteria
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

4. Secondary Outcome: Efficacy, as Assessed by Proportion of Assessments With 1-grade Improvement, Using West Haven Criteria
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy, as Assessed by Time Spent in an Improved State by 1 or 2 Grades Using the West Haven Criteria
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

6. Secondary Outcome: Efficacy, as Assessed by Percentage of Subjects With a 1 or 2 Grade Improvement, Using the West Haven Criteria
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 96 hours
Reporting Status: Not Posted

7. Secondary Outcome: Efficacy, as Assessed by Severity of Hepatic Encephalopathy Using the Glasgow Coma Scale
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

8. Secondary Outcome: Effects of Ammonul® on Blood Ammonia Levels, Amino Acids and Carnitine
Time Frame: 96 hours of treatment and follow-up
Reporting Status: Not Posted

9. Secondary Outcome: Pharmacokinetic Characteristics of Ammonul® and Its Metabolites
Time Frame: Every 24 hours during treatment period of 96 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No information available.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One participant was enrolled but did not receive drug or was randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other